CLINICAL TRIAL: NCT00713934
Title: Autologous Transplantation of Bone Marrow Derived CD 133 Positive Stem Cell and Mono Nuclear Cell (MNC) Transplantation in Patients With Decompensate Cirrhosis: Randomized Clinical Trial
Brief Title: Autologous Bone Marrow Stem Cells in Cirrhosis Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Collaborators: Small Business Developing Center (Unknown); Shiraz University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Liver-001
Record Dates: First submitted 2008-07-09; First posted 2008-07-14 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2010-03

CONDITIONS: Stem Cell Transplantation; Cirrhosis
Keywords: Autologous Bone marrow stem cells; Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: CD133
- 2 (Experimental)
  Interventions: Biological: BM-MNC

INTERVENTIONS:
Biological: CD133 — portal vein infusion of CD133+ cells
  Arms: 1
Biological: BM-MNC — portal vein infusion of BM-MNC
  Arms: 2

SUMMARY:
Liver cirrhosis (LC) is the end stage of chronic liver disease. The liver transplantation is one of the only effective therapies available to such patients. However, lack of donors, surgical complications, rejection, and high cost are it's serious problems. The potential for stem cells in bone marrow (BM) to differentiate into hepatocytes cells was recently confirmed. Moreover, BMC transplantation has been performed to treat hematological diseases, and several clinical studies have applied BMC injection to induce regeneration of myocardium and blood vessels. In this study we will evaluate safety and feasibility of autologous bone marrow mono nuclear (BM-MNC) and enriched CD133+ hematopoietic stem cell transplantation through the portal vein in patients with decompensate cirrhosis.

DETAILED DESCRIPTION:
BM (200 ml) will be harvested from the iliac crest according to standard procedures under general anesthesia and is collected in plastic bags containing anti coagulant. After precipitation of red blood cells, Low density mononuclear cells will be collected by centrifugation in Ficoll-Paque density gradient. For CD133+ cells separation the CliniMACS instrument will be used. Cells are injected via portal vein under sonography monitoring. After cell therapy, patients are followed up every week for 4 weeks, and laboratory data are analyzed for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Liver biopsy showing histological Cirrhosis, grade B or C (Child-Pugh score)
* Alkaline phosphatase between 2 X to 3X normal value
* liver Cirrhosis in Sonography study
* Incomplete response to UDCA after 6 months of treatment.
* Negative pregnancy test (female patients in fertile age)
* written consent

Exclusion Criteria:

* Presence of active hepatic encephalopathy
* Refractory ascites
* Evidences of active autoimmune liver disease (e.g. gamma globulin of more than 2 times of upper limit of normal, and ALT > 3 times normal in patients with autoimmune hepatitis)
* Hepatocellular carcinoma or other malignancies
* sepsis
* Presence of significant extrahepatic biliary disease (e.g. CBD stone, PSC, etc.)
* HIV, HBV or HCV infection
* Cardiac, renal or respiratory failure
* Active thrombosis of the portal or hepatic veins
* INR>2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Liver function test | 6 months
MELD score | 6 months

SECONDARY OUTCOMES:
Cirrhosis mortality | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gorabi, PhD, Study Chair — Royan institute, Tehran, Iran; Malekhosseini, MD, Study Chair — Liver Transplantation Research Center, Shiraz, Iran; Hossein Baharvand, PhD, Principal Investigator — Royan institute, Tehran, Iran; Saman Nikeghbal, MD, Principal Investigator — Liver Transplantation Research Center, Shiraz, Iran; Nasser Aghdami, MD, PhD, Study Director — Royan institute, Tehran, Iran
Locations (2):
- Iran (2):
  - Liver Transplant Research Center, Shiraz, Fars
  - Royan Institute, Tehran, Tehran Province

REFERENCES:
- [Derived] Nikeghbalian S, Pournasr B, Aghdami N, Rasekhi A, Geramizadeh B, Hosseini Asl SM, Ramzi M, Kakaei F, Namiri M, Malekzadeh R, Vosough Dizaj A, Malek-Hosseini SA, Baharvand H. Autologous transplantation of bone marrow-derived mononuclear and CD133(+) cells in patients with decompensated cirrhosis. Arch Iran Med. 2011 Jan;14(1):12-7. PMID 21194255
- See also: Royan Institute — http://www.royaninstitute.org